CLINICAL TRIAL: NCT02080728
Title: Transversus Abdominis Plane Block During Kidney Transplant Surgery: Prospective Controlled Randomized Double-blind Trial Comparing Ropivacaine 0.2% With Placebo.
Brief Title: Transversus Abdominis Plane Block During Kidney Transplant Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Jazayeri-Steinmetz AOI 2012
Record Dates: First submitted 2014-03-05; First posted 2014-03-06 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Kidney Transplant
MeSH Terms: interventions — Ropivacaine

ARMS (2):
- TAP-Bloc (Experimental)
  Interventions: Drug: Ropivacaine 500mg/100ml Naropeine
- Control (Placebo Comparator)
  Interventions: Drug: 0.9% sodium chloride BAXTER

INTERVENTIONS:
Drug: Ropivacaine 500mg/100ml Naropeine
  Arms: TAP-Bloc
Drug: 0.9% sodium chloride BAXTER
  Arms: Control

SUMMARY:
The surgeon places the catheter in the thickness of the oblique internal and transverse muscles at the moment the wall is closed, under visual control. A multiperforated catheter whose length corresponds to that of the incision is chosed. The catheter will deliver one of two products chosen at random: either ropivacaine or placebo.

This study will evaluate postoperative pain during the first 24 hours thanks to a recognized indicator the VAS (Visual Analogue pain Scale). The total consumption of analgesics will also be recorded, starting with the titration of morphine in the post-op room, and then the consumption of classical analgesics in the nephrology department. These will only be given if the VAS score is equal to 4 or above.

This is a prospective, single-centre, controlled, double blind study of ropivacaïne 0.2% versus placebo in continuous TAP block during the first 24 hours after the operation in patients undergoing kidney transplant surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient opéré for kidney transplant
* Patients who have provided written informed consent
* Patients with national health insurance cover
* Patients aged 18 years and above

Exclusion Criteria:

* Pregnant or breast-feeding women
* allergies/hypersensitivity to paracetamol (or propacetamol chlorhydrate (paracetamol pro-drug) or one of its excipients), to local anesthetics, morphines (or other constituents)
* patients under guardianship or ward of court

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07-23 (Actual); Primary Completion 2014-07-09 (Actual); Study Completion 2014-07-09 (Actual)

PRIMARY OUTCOMES:
Mesurement of VAS (Visual analogue scale) scores for pain | During the first 24 hours post-op

SECONDARY OUTCOMES:
Measurement of analgesic consomption | During the first 24 hours post-op

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France